CLINICAL TRIAL: NCT06207266
Title: A Prospective Study of the Impact of an Emotional Intelligence Program on Opioid Relapse and Its Determinants
Brief Title: Impact Emotional Intelligence Program on Opioid Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, lecturer of psychiatry, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EMOTION INTELLIGENCE
Record Dates: First submitted 2023-12-17; First posted 2024-01-16 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Emotional Intelligence; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants with opioid use disorder were divided into two groups: group with emotion intelligence program (n=20) and group without intelligence program (n=20). A healthy group (n=20) served as a control group.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participants with opioid use disorder group with emotion intelligence program (n=20) (Experimental): Participants with opioid use disorder group who had emotion intelligence program to increase aware about definition, component, how to deal with EI to reduce relapse rate.
  Interventions: Behavioral: emotion intelligence program
- Participants with opioid use disorder group without intelligence program (n=20). (No Intervention): Participants with opioid use disorder group who had traditional medical treatment only
- A healthy group (n=20) served as a control group. (No Intervention): A healthy group who did not have history of psychiatric illness or substance use.

INTERVENTIONS:
Behavioral: emotion intelligence program — The programme was established using research that described emotional intelligence components and their applicability to patients suffering from substance abuse. it considers as awareness program.
  Arms: Participants with opioid use disorder group with emotion intelligence program (n=20)

SUMMARY:
Addiction is the repeated and increased use of a substance, the deprivation of which gives rise to symptoms of distress and an irresistible urge to use the agent again and which leads also to physical and mental deterioration. The concept of emotional intelligent (EI) "the ability to perceive accurately, appraise and express emotion; the ability to access and generate feelings when they facilitate thought; the ability to understand emotion and emotional knowledge; and the ability to regulate emotions to promote emotional and intellectual growth". Most drug addicts possess hidden defects in their social skills, and do not have good relations with their peers.

DETAILED DESCRIPTION:
Addiction is the repeated and increased use of a substance, the deprivation of which gives rise to symptoms of distress and an irresistible urge to use the agent again and which leads also to physical and mental deterioration. Continued opioid misuse can result in syndromes of abuse and dependence and cause disturbances in mood, behavior, and cognition that can mimic other psychiatric disorders. Opioid addiction affects the young and the old, the wealthy and the poor, and the professional and the unemployed.

The concept of emotional intelligent (EI) "the ability to perceive accurately, appraise and express emotion; the ability to access and generate feelings when they facilitate thought; the ability to understand emotion and emotional knowledge; and the ability to regulate emotions to promote emotional and intellectual growth", the ability to manage and regulate emotions in an effective manner and ability to be sufficiently optimistic, positive and self- motivated in order to set and achieve goals.

Most drug addicts possess hidden defects in their social skills, and do not have good relations with their peers. The other possible causes of orienting toward drugs are defects in problem solving, stress-management, and prevention from dangerous and impulsive behaviors.

ELIGIBILITY:
Inclusion Criteria:

* in opioid groups: only opioid addiction
* in healthy groups: no history of psychiatric illness or substance use

Exclusion Criteria:

* have medical conditions

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
measure level of emotion intelligence in opioid addiction | through study completion, an average of 1 year
  Measure the level of emotional intelligence. The scale consists of sixty objects classified into six distinct domains. A four-point Likert scale is employed, which spans from 1 (indicating never) to 4 (indicating always). The percentages represent the scores; emotional intelligence ranges (from 0-100%), and higher scores mean a high level of emotional intelligence.
develop an EI programme to prevent relapses in addiction. | through study completion, an average of 1 year
  An emotional intelligence (EI) program was developed and implemented for patients in the hospital. Emotion intelligence scale was measured at baseline prior to starting the EI program. The EI program was then administered to patients during their hospital stay. Emotion intelligence scale assessments were conducted at discharge from the hospital and again 3 months after discharge. Regarding EI program sessions took place in the recreation hall, where material such as videos and booklets containing content on emotional intelligence skills was presented.

CONTACTS AND LOCATIONS:
Overall Officials: gellan Karamallah R Ahmed, Study Director — Assiut University
Locations (1):
- Faculty of Nursing, Asyut, Egypt